CLINICAL TRIAL: NCT03003559
Title: Comparison of High Flow Nasal Cannula vs Nasal Cannula in Mild Chronic Obstructive Pulmonary Disease Exacerbation(AECOPD)
Brief Title: HFNC vs Nasal Cannula in Mild Chronic Obstructive Pulmonary Disease Exacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Qingyuan Zhan, head of Pulmonary and Critical care medicine ward 4, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1304304-1
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: COPD Exacerbation
Keywords: COPD Exacerbation; High Flow Oxygen; Nasal Cannula; mild
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flow nasal cannula (Experimental): High flow nasal cannula(OptiflowTM); Flow 25-60 L/min is set according to patients' comfort; FiO2 is adjusted to maintain peripheral capillary oxygen saturation(SpO2) 90-95%; temperature is set at 37.
  Interventions: Device: High flow nasal cannula
- Nasal cannula (No Intervention): Nasal cannula;set oxygen flow to keep SpO2 90-95%

INTERVENTIONS:
Device: High flow nasal cannula — High flow nasal cannula (HFNC) is a new emerging noninvasive respiratory support technology, which mainly includes high flow (15-60 L/min) device, heating humidification device and nasal cannula for high flow. A large number of physiological studies confirmed that HFNC has the following critical physiological effects: promoting airway humidification, improving tolerance of treatment, reducing the physiological dead space on the upper respiratory tract, producing a certain level of positive end expiratory pressure (2-7 cmH2O), decreasing the work of breathing and so on.
  Other Names: High flow oxygen
  Arms: High flow nasal cannula

SUMMARY:
For AECOPD patients, only 8% patients ventilated by noninvasive and invasive positive pressure ventilation. Nasal cannula is the most common pattern of oxygen therapy in mild AECOPD. As a low flow oxygen therapy, nasal cannula has many disadvantages.Therefore, we design a randomized controlled trial(RCT)to explore whether HFNC would be better than nasal cannula to prevent the aggravation of respiratory failure and endotracheal intubation in mild AECOPD.

DETAILED DESCRIPTION:
For AECOPD patients, most of patients don't need respiratory support, only 8% patients ventilated by noninvasive and invasive positive pressure ventilation. Nasal cannula is the most common pattern of oxygen therapy in mild AECOPD. As a low flow oxygen therapy, nasal cannula has many disadvantages: discomfort, low humidity and unstable fraction of inspired oxygen(FiO2) in inspiratory gas. Therefore, we design a RCT to explore whether HFNC would be better than nasal cannula to prevent the aggravation of respiratory failure and endotracheal intubation in mild AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD; pH≥7.35, PaCO2>45 mmHg

Exclusion Criteria:

* Need to be intubated immediately; refuse to engage in the study; severe organ dysfunction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
endotracheal intubation demand rate | 90days

SECONDARY OUTCOMES:
actual endotracheal intubation rate | 90days

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhan, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia J, Yang H, Zhan Q, Fan Y, Wang C. High-flow nasal cannula may prolong the length of hospital stay in patients with hypercapnic acute COPD exacerbation. Respir Med. 2023 Dec;220:107465. doi: 10.1016/j.rmed.2023.107465. Epub 2023 Nov 11. PMID 37956934
- [Derived] Xia J, Gu S, Lei W, Zhang J, Wei H, Liu C, Zhang H, Lu R, Zhang L, Jiang M, Hu C, Cheng Z, Wei C, Chen Y, Lu F, Chen M, Bi H, Liu H, Yan C, Teng H, Yang Y, Liang C, Ge Y, Hou P, Liu J, Gao W, Zhang Y, Feng Y, Tao C, Huang X, Pan P, Luo H, Yun C, Zhan Q. High-flow nasal cannula versus conventional oxygen therapy in acute COPD exacerbation with mild hypercapnia: a multicenter randomized controlled trial. Crit Care. 2022 Apr 15;26(1):109. doi: 10.1186/s13054-022-03973-7. PMID 35428349